CLINICAL TRIAL: NCT06275789
Title: Mix of Demineralized Freeze-Dried Bone Allograft and Deproteinized Bovine Bone Mineral: a Possible Solution for Alveolar Ridge Preservation?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: Geistlich Pharma AG (Industry); ZimVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-268
Record Dates: First submitted 2024-02-07; First posted 2024-02-23 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Alveolar Ridge Preservation; Dental Extraction; Bone Graft

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test Group (Experimental): This group will receive the grafting material that is a combination of DFDBA + DBBM + collagen matrix seal during the alveolar ridge preservation procedure.
  Interventions: Procedure: Alveolar ridge preservation
- Control Group (Active Comparator): This group will receive the grafting material that is a Tutoplast® processed mineralized particulate allograft + collagen matrix seal during the alveolar ridge preservation procedure.
  Interventions: Procedure: Alveolar ridge preservation

INTERVENTIONS:
Procedure: Alveolar ridge preservation — Premolar tooth will be extracted flapless and ridge preservation procedure with bone grafting material will be done.

SUMMARY:
The purpose of the study is to compare a new grafting material for alveolar ridge preservation to a commonly used and well studied material. Alveolar ridge dimensions as well as histology will be compared.

DETAILED DESCRIPTION:
Brief Background and Goal: Dimensional changes following extractions are inevitable. Many techniques and combinations of materials have been studied and shown to be effective at minimizing these changes. Although no material has been able to fully preserve the ridge, xenografts have been shown to be the most effective at maintaining the volume, however, the use of demineralized freeze-dried bone allograft (DFDBA) results in the most vital bone when evaluated histologically. These factors are important when planning for a successful future implant supported prosthesis. A new material that combines xenograft (deproteinized bovine bone mineral - DBBM) with DFDBA has recently been introduced to the market. The aim of the study is to compare the dimensional and histological changes following flapless alveolar ridge preservation (ARP) in the premolar and molar region with a new material that combines DFDBA and DBBM to a commonly used mineralized allograft.

Research Question: In patients who require an extraction for future implant placement, during alveolar ridge preservation, will combining demineralized freeze-dried bone allograft (DFDBA) and deproteinized bovine bone mineral (DBBM) compared to Tutoplast® processed mineralized particulate allograft result in less dimensional changes at the time of implant placement 4 months later.

Specific Aims: The primary goal of the study is to compare the dimensional changes following alveolar ridge preservation with a new material that combines DFDBA and DBBM to a commonly used mineralized allograft material. The secondary goal is to assess the histological composition of the bone after 4 months of healing. The additional goals are to measure possible confounding factors on the dimensional changes of the alveolar ridge.

Significance: The goal behind the combination of DBBM and DFDBA is to evaluate whether there could potentially be a synergistic effect between the two materials that would make it a more desirable material to use for ARP procedures.

Innovation: There is currently no published research that compares the combination of DFDBA and DBBM to a conventional method inside the extraction site during an alveolar ridge preservation procedure. This grafting material is new on the market and the first of its kind.

Research Plan: The randomized clinical trial will be performed at the Nova Southeastern College of Dental Medicine in the Post-graduate Periodontology Clinic. 30 patients requiring premolar or molar extraction with future implant placement will be randomly divided into 2 groups, one test and one control. Following extraction, the patients will receive either allograft or graft combination of DFDBA and DBBM. The changes in horizontal and vertical dimensions of the alveolar ridge as well as the histology will be assessed and compared at 4 months.

Expected Results: When compared to allograft, the graft mixture containing the DFDBA and DBBM will maintain greater dimensional volume due to the dimensionally stable properties of DBBM and will contain more vital bone due to the osteoinductive properties of DFDBA.

ELIGIBILITY:
Inclusion Criteria:

* Patients in good health
* Require the extraction of at least one premolar or molar with future implant placement
* Sufficient keratinized gingiva (equal or more than 2mm prior to extraction),
* No more than 3mm of buccal bone loss
* Flapless extraction possible
* Full mouth plaque index of less than 25%

Exclusion Criteria:

* Nicotine consumption equivalent to or more than 10 cigarettes per day
* Electronic cigarette usage
* A history of irradiation of head and neck area
* Immunodeficiency disease
* Uncontrolled systemic health problems (hypertension crisis 180/120, hyperthyroidism, diabetes with HbA1c over 7, recent history of stroke, cancer) History of medications that affect bone remodeling process (bisphosphonates, RANK-L inhibitors)
* Previous adverse reaction to the biomaterials used
* Pregnancy/lactation, or those who are trying to become pregnant.
* Active uncontrolled or untreated periodontal disease
* Periapical lesions greater than 1 cm and soft tissue pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
changes in horizontal dimensions of the alveolar ridge | 4 months
  Soft and hard tissue horizontal dimensions of the alveolar ridge will be measured after extraction and 4 months later.
changes in vertical dimensions of the alveolar ridge | 4 months
  Soft and hard tissue vertical dimensions of the alveolar ridge will be measured after extraction and 4 months later.

SECONDARY OUTCOMES:
vital bone percentage | 4 months
  vital bone percentage will evaluated histologically following biopsy at time of implant placement.

OTHER OUTCOMES:
thickness of the buccal plate in mm and its influence on the ridge dimension | 4 months
  the thickness of the buccal plate will be measured digitally to assess if it may be a confounding factor
the thickness of the lingual plate in mm and its influence on the ridge dimension | 4 months
  the thickness of the lingual plate will be measured digitally to assess if it may be a confounding factor
the thickness of the overlying buccal soft tissue in mm and its influence on the ridge dimension | 4 months, 1 year
  the thickness of the overlying soft tissue will be measured digitally to assess if it may be a confounding factor
the position of extraction site (maxilla vs. mandible) and its influence on the ridge dimension | 4 months, 1 year
  the position of the tooth in the arch will be analyzed to assess if it may be a confounding factor
# of cigarettes and its influence on the ridge dimension | 4 months
  the quantity of cigarettes will be analyzed to assess if it may be a confounding factor
oral hygiene using the plaque index and its influence on the ridge dimension | 4 months, 1 year
  the effectiveness of oral hygiene will be analyzed to assess if it may be a confounding factor

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Southeastern University, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amler MH. The time sequence of tissue regeneration in human extraction wounds. Oral Surg Oral Med Oral Pathol. 1969 Mar;27(3):309-18. doi: 10.1016/0030-4220(69)90357-0. No abstract available. PMID 5251474
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Background] Buser D, Chappuis V, Belser UC, Chen S. Implant placement post extraction in esthetic single tooth sites: when immediate, when early, when late? Periodontol 2000. 2017 Feb;73(1):84-102. doi: 10.1111/prd.12170. PMID 28000278
- [Background] Tan WL, Wong TL, Wong MC, Lang NP. A systematic review of post-extractional alveolar hard and soft tissue dimensional changes in humans. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:1-21. doi: 10.1111/j.1600-0501.2011.02375.x. PMID 22211303
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Hammerle CH, Chen ST, Wilson TG Jr. Consensus statements and recommended clinical procedures regarding the placement of implants in extraction sockets. Int J Oral Maxillofac Implants. 2004;19 Suppl:26-8. No abstract available. PMID 15635943
- [Background] Ten Heggeler JM, Slot DE, Van der Weijden GA. Effect of socket preservation therapies following tooth extraction in non-molar regions in humans: a systematic review. Clin Oral Implants Res. 2011 Aug;22(8):779-88. doi: 10.1111/j.1600-0501.2010.02064.x. Epub 2010 Nov 22. PMID 21091540
- [Background] Avila-Ortiz G, Gubler M, Romero-Bustillos M, Nicholas CL, Zimmerman MB, Barwacz CA. Efficacy of Alveolar Ridge Preservation: A Randomized Controlled Trial. J Dent Res. 2020 Apr;99(4):402-409. doi: 10.1177/0022034520905660. Epub 2020 Feb 12. PMID 32050833
- [Background] Abellan D, Barallat L, Vilarrasa J, Cabezas M, Pascual La Rocca A, Valles C, Nart J. Ridge preservation in molar sites comparing xenograft versus mineralized freeze-dried bone allograft: A randomized clinical trial. Clin Oral Implants Res. 2022 May;33(5):511-523. doi: 10.1111/clr.13911. Epub 2022 Mar 14. PMID 35218248
- [Background] Buser D, Martin W, Belser UC. Optimizing esthetics for implant restorations in the anterior maxilla: anatomic and surgical considerations. Int J Oral Maxillofac Implants. 2004;19 Suppl:43-61. PMID 15635945
- [Background] Canullo L, Tallarico M, Radovanovic S, Delibasic B, Covani U, Rakic M. Distinguishing predictive profiles for patient-based risk assessment and diagnostics of plaque induced, surgically and prosthetically triggered peri-implantitis. Clin Oral Implants Res. 2016 Oct;27(10):1243-1250. doi: 10.1111/clr.12738. Epub 2015 Nov 20. PMID 26584716
- [Background] Evans CD, Chen ST. Esthetic outcomes of immediate implant placements. Clin Oral Implants Res. 2008 Jan;19(1):73-80. doi: 10.1111/j.1600-0501.2007.01413.x. Epub 2007 Oct 22. PMID 17956569
- [Background] Araujo MG, Sukekava F, Wennstrom JL, Lindhe J. Ridge alterations following implant placement in fresh extraction sockets: an experimental study in the dog. J Clin Periodontol. 2005 Jun;32(6):645-52. doi: 10.1111/j.1600-051X.2005.00726.x. PMID 15882225
- [Background] Avila-Ortiz G, Chambrone L, Vignoletti F. Effect of alveolar ridge preservation interventions following tooth extraction: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:195-223. doi: 10.1111/jcpe.13057. Erratum In: J Clin Periodontol. 2020 Jan;47(1):129. doi: 10.1111/jcpe.13212. PMID 30623987
- [Background] Avila-Ortiz G, Elangovan S, Kramer KW, Blanchette D, Dawson DV. Effect of alveolar ridge preservation after tooth extraction: a systematic review and meta-analysis. J Dent Res. 2014 Oct;93(10):950-8. doi: 10.1177/0022034514541127. Epub 2014 Jun 25. PMID 24966231
- [Background] Darby I, Chen ST, Buser D. Ridge preservation techniques for implant therapy. Int J Oral Maxillofac Implants. 2009;24 Suppl:260-71. PMID 19885449
- [Background] Khan SN, Cammisa FP Jr, Sandhu HS, Diwan AD, Girardi FP, Lane JM. The biology of bone grafting. J Am Acad Orthop Surg. 2005 Jan-Feb;13(1):77-86. PMID 15712985
- [Background] Aladmawy MA, Natto ZS, Kreitzer M, Ogata Y, Hur Y. Histological and histomorphometric evaluation of alveolar ridge preservation using an allograft and nonresorbable membrane with and without primary closure: A pilot randomized controlled clinical trial. Medicine (Baltimore). 2022 Jul 1;101(26):e29769. doi: 10.1097/MD.0000000000029769. PMID 35777057
- [Background] Borg TD, Mealey BL. Histologic healing following tooth extraction with ridge preservation using mineralized versus combined mineralized-demineralized freeze-dried bone allograft: a randomized controlled clinical trial. J Periodontol. 2015 Mar;86(3):348-55. doi: 10.1902/jop.2014.140483. Epub 2014 Nov 21. PMID 25415247
- [Background] Brugnami F, Then PR, Moroi H, Leone CW. Histologic evaluation of human extraction sockets treated with demineralized freeze-dried bone allograft (DFDBA) and cell occlusive membrane. J Periodontol. 1996 Aug;67(8):821-5. doi: 10.1902/jop.1996.67.8.821. PMID 8866322
- [Background] Canullo L, Del Fabbro M, Khijmatgar S, Panda S, Ravida A, Tommasato G, Sculean A, Pesce P. Dimensional and histomorphometric evaluation of biomaterials used for alveolar ridge preservation: a systematic review and network meta-analysis. Clin Oral Investig. 2022 Jan;26(1):141-158. doi: 10.1007/s00784-021-04248-1. Epub 2021 Nov 26. PMID 34826029
- [Background] Cardaropoli D, Tamagnone L, Roffredo A, Gaveglio L, Cardaropoli G. Socket preservation using bovine bone mineral and collagen membrane: a randomized controlled clinical trial with histologic analysis. Int J Periodontics Restorative Dent. 2012 Aug;32(4):421-30. PMID 22577648
- [Background] Chan HL, Lin GH, Fu JH, Wang HL. Alterations in bone quality after socket preservation with grafting materials: a systematic review. Int J Oral Maxillofac Implants. 2013 May-Jun;28(3):710-20. doi: 10.11607/jomi.2913. PMID 23748301
- [Background] Corning PJ, Mealey BL. Ridge preservation following tooth extraction using mineralized freeze-dried bone allograft compared to mineralized solvent-dehydrated bone allograft: A randomized controlled clinical trial. J Periodontol. 2019 Feb;90(2):126-133. doi: 10.1002/JPER.18-0199. Epub 2018 Sep 19. PMID 30161278
- [Background] De Risi V, Clementini M, Vittorini G, Mannocci A, De Sanctis M. Alveolar ridge preservation techniques: a systematic review and meta-analysis of histological and histomorphometrical data. Clin Oral Implants Res. 2015 Jan;26(1):50-68. doi: 10.1111/clr.12288. Epub 2013 Nov 1. PMID 27007188
- [Background] Demetter RS, Calahan BG, Mealey BL. Histologic Evaluation of Wound Healing After Ridge Preservation With Cortical, Cancellous, and Combined Cortico-Cancellous Freeze-Dried Bone Allograft: A Randomized Controlled Clinical Trial. J Periodontol. 2017 Sep;88(9):860-868. doi: 10.1902/jop.2017.170155. Epub 2017 Apr 28. PMID 28452622
- [Background] Eskow AJ, Mealey BL. Evaluation of healing following tooth extraction with ridge preservation using cortical versus cancellous freeze-dried bone allograft. J Periodontol. 2014 Apr;85(4):514-24. doi: 10.1902/jop.2013.130178. Epub 2013 May 31. PMID 23725026
- [Background] Froum S, Cho SC, Rosenberg E, Rohrer M, Tarnow D. Histological comparison of healing extraction sockets implanted with bioactive glass or demineralized freeze-dried bone allograft: a pilot study. J Periodontol. 2002 Jan;73(1):94-102. doi: 10.1902/jop.2002.73.1.94. PMID 11846205
- [Background] Iasella JM, Greenwell H, Miller RL, Hill M, Drisko C, Bohra AA, Scheetz JP. Ridge preservation with freeze-dried bone allograft and a collagen membrane compared to extraction alone for implant site development: a clinical and histologic study in humans. J Periodontol. 2003 Jul;74(7):990-9. doi: 10.1902/jop.2003.74.7.990. PMID 12931761
- [Background] Nelson AC, Mealey BL. A randomized controlled trial on the impact of healing time on wound healing following ridge preservation using a 70%/30% combination of mineralized and demineralized freeze-dried bone allograft. J Periodontol. 2020 Oct;91(10):1256-1263. doi: 10.1002/JPER.19-0610. Epub 2020 Mar 3. PMID 32052432
- [Background] Poulias E, Greenwell H, Hill M, Morton D, Vidal R, Shumway B, Peterson TL. Ridge preservation comparing socket allograft alone to socket allograft plus facial overlay xenograft: a clinical and histologic study in humans. J Periodontol. 2013 Nov;84(11):1567-75. doi: 10.1902/jop.2013.120585. Epub 2013 Jan 23. PMID 23339378
- [Background] Sadeghi R, Babaei M, Miremadi SA, Abbas FM. A randomized controlled evaluation of alveolar ridge preservation following tooth extraction using deproteinized bovine bone mineral and demineralized freeze-dried bone allograft. Dent Res J (Isfahan). 2016 Mar-Apr;13(2):151-9. doi: 10.4103/1735-3327.178202. PMID 27076830
- [Background] Saito H, Couso-Queiruga E, Shiau HJ, Stuhr S, Prasad H, Allareddy TV, Reynolds MA, Avila-Ortiz G. Evaluation of poly lactic-co-glycolic acid-coated beta-tricalcium phosphate for alveolar ridge preservation: A multicenter randomized controlled trial. J Periodontol. 2021 Apr;92(4):524-535. doi: 10.1002/JPER.20-0360. Epub 2020 Oct 12. PMID 32996128
- [Background] Scheyer ET, Heard R, Janakievski J, Mandelaris G, Nevins ML, Pickering SR, Richardson CR, Pope B, Toback G, Velasquez D, Nagursky H. A randomized, controlled, multicentre clinical trial of post-extraction alveolar ridge preservation. J Clin Periodontol. 2016 Dec;43(12):1188-1199. doi: 10.1111/jcpe.12623. Epub 2016 Oct 21. PMID 27617409
- [Background] Serrano Mendez CA, Lang NP, Caneva M, Ramirez Lemus G, Mora Solano G, Botticelli D. Comparison of allografts and xenografts used for alveolar ridge preservation. A clinical and histomorphometric RCT in humans. Clin Implant Dent Relat Res. 2017 Aug;19(4):608-615. doi: 10.1111/cid.12490. Epub 2017 May 2. PMID 28466494
- [Background] Suarez-Lopez Del Amo F, Monje A. Efficacy of biologics for alveolar ridge preservation/reconstruction and implant site development: An American Academy of Periodontology best evidence systematic review. J Periodontol. 2022 Dec;93(12):1827-1847. doi: 10.1002/JPER.22-0069. Epub 2022 Oct 24. PMID 35841608
- [Background] Toloue SM, Chesnoiu-Matei I, Blanchard SB. A clinical and histomorphometric study of calcium sulfate compared with freeze-dried bone allograft for alveolar ridge preservation. J Periodontol. 2012 Jul;83(7):847-55. doi: 10.1902/jop.2011.110470. Epub 2011 Dec 13. PMID 22166162
- [Background] Wang HL, Tsao YP. Histologic evaluation of socket augmentation with mineralized human allograft. Int J Periodontics Restorative Dent. 2008 Jun;28(3):231-7. PMID 18605598
- [Background] Whetman J, Mealey BL. Effect of Healing Time on New Bone Formation After Tooth Extraction and Ridge Preservation With Demineralized Freeze-Dried Bone Allograft: A Randomized Controlled Clinical Trial. J Periodontol. 2016 Sep;87(9):1022-9. doi: 10.1902/jop.2016.160139. Epub 2016 Apr 30. PMID 27133791
- [Background] Wood RA, Mealey BL. Histologic comparison of healing after tooth extraction with ridge preservation using mineralized versus demineralized freeze-dried bone allograft. J Periodontol. 2012 Mar;83(3):329-36. doi: 10.1902/jop.2011.110270. Epub 2011 Jul 12. PMID 21749166
- [Background] Zampara E, Alshammari M, De Bortoli J, Mullings O, Gkisakis IG, Benalcazar Jalkh EB, Tovar N, Coelho PG, Witek L. A Histologic and Histomorphometric Evaluation of an Allograft, Xenograft, and Alloplast Graft for Alveolar Ridge Preservation in Humans: A Randomized Controlled Clinical Trial. J Oral Implantol. 2022 Dec 1;48(6):541-549. doi: 10.1563/aaid-joi-D-21-00012. PMID 35446950
- [Background] Zellner JW, Allen HT, Kotsakis GA, Mealey BL. Wound healing after ridge preservation: A randomized controlled trial on short-term (4 months) versus long-term (12 months) histologic outcomes. J Periodontol. 2023 May;94(5):622-629. doi: 10.1002/JPER.22-0187. Epub 2023 Jan 10. PMID 36527199
- [Background] Canellas JVDS, Soares BN, Ritto FG, Vettore MV, Vidigal Junior GM, Fischer RG, Medeiros PJD. What grafting materials produce greater alveolar ridge preservation after tooth extraction? A systematic review and network meta-analysis. J Craniomaxillofac Surg. 2021 Nov;49(11):1064-1071. doi: 10.1016/j.jcms.2021.06.005. Epub 2021 Jun 19. PMID 34176715
- [Background] Mayer Y, Ginesin O, Zigdon-Giladi H. Socket Preservation Using Xenograft Does Not Impair Implant Primary Stability in Sheep: Clinical, Histological, and Histomorphometric Study. J Oral Implantol. 2020 Dec 1;46(6):580-588. doi: 10.1563/aaid-joi-D-19-00237. PMID 32315436
- [Background] Monje A, Ravida A, Wang HL, Helms JA, Brunski JB. Relationship Between Primary/Mechanical and Secondary/Biological Implant Stability. Int J Oral Maxillofac Implants. 2019 Suppl;34:s7-s23. doi: 10.11607/jomi.19suppl.g1. PMID 31116830